CLINICAL TRIAL: NCT06999746
Title: Effectiveness of Using Force Sensing Resistor to Assist Oropharyngeal Rehabilitation in Patients With Obstructive Sleep Apnea Using Continuous Positive Airway Pressure
Brief Title: Device-Assisted Oropharyngeal Rehabilitation in Obstructive Sleep Apnea Patients Using Continuous Positive Airway Pressure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-113-050
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sleep hygiene education (Sham Comparator): Receive monthly sleep hygiene education
  Interventions: Other: Control
- Oropharyngeal rehabilitation (Experimental): Receive oropharyngeal rehabilitation training over three months
  Interventions: Device: Oropharyngeal Exercise
- Continuous positive airway pressure (Experimental): Receive continuous positive airway pressure
  Interventions: Device: Continuous positive airway pressure
- Continuous positive airway pressure and oropharyngeal rehabilitation (Experimental): Receive continuous positive airway pressure and oropharyngeal rehabilitation training for three months
  Interventions: Device: Continuous positive airway pressure and oropharyngeal exercise

INTERVENTIONS:
Other: Control — Sleep hygiene education
  Arms: Sleep hygiene education
Device: Oropharyngeal Exercise — Device-monitoring oropharyngeal exercise, 1-5 days a week for three months
  Arms: Oropharyngeal rehabilitation
Device: Continuous positive airway pressure — Continuous positive airway pressure, 1-5 days a week for three months
  Arms: Continuous positive airway pressure
Device: Continuous positive airway pressure and oropharyngeal exercise — Continuous positive airway pressure and device-monitoring oropharyngeal exercise, 1-5 days a week for three months
  Arms: Continuous positive airway pressure and oropharyngeal rehabilitation

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of device-assisted oropharyngeal rehabilitation (OPR) in improving upper airway muscle function and reducing obstructive sleep apnea (OSA) severity in adult patients diagnosed with OSA who are receiving continuous positive airway pressure (CPAP) therapy.

The main questions it aims to answer are:

1. Does combining OPR with CPAP increase upper airway space volume compared to using CPAP alone?
2. Does OPR improve tongue muscle strength, and is this improvement associated with reduced CPAP pressure requirements?
3. Do patients receiving OPR (alone or combined with CPAP) show greater improvements in OSA severity and clinical symptoms compared to those receiving CPAP alone or no intervention? Researchers will compare four groups-Control, OPR-only, CPAP-only, and CPAP + OPR-to see if device-assisted OPR enhances treatment outcomes beyond CPAP alone.

Participants will:

1. Be randomly assigned to one of four groups (Control, OPR-only, CPAP-only, CPAP+OPR).
2. Perform home-based OPR exercises (30-45 minutes/session, 1-2 sessions/day, 3-5 days/week for 3 months) in the OPR and CPAP+OPR groups.
3. Have their exercise monitored using a strength sensor, with intensity adjusted every 2-4 weeks during hospital visits.
4. Undergo assessments before and after the intervention, including:

(1) Polysomnography for OSA severity, (2) CT and ultrasound for upper airway and tongue muscle structure, (3) Tongue muscle strength/endurance tests, (4) Sleep quality questionnaires, (5) CPAP usage and pressure reports.

DETAILED DESCRIPTION:
Background: Obstructive sleep apnea (OSA) is a common respiratory disorder associated with various complications, including cardiovascular, metabolic, and cognitive issues. Continuous positive airway pressure (CPAP) therapy can effectively reduce sleep apnea events and decrease the incidence of related complications. However, studies have shown that approximately half of OSA patients attempting CPAP therapy either cannot tolerate CPAP at all or only partially comply with it. Oropharyngeal rehabilitation (OPR), which involves isometric and isotonic exercises, can enhance the muscle tone of the tongue, pharynx, and soft palate. OPR may serve as one of the treatment options for OSA. Nevertheless, there is limited literature exploring the combined treatment approach of CPAP and OPR.

Methods：This study will recruit 30 200 adult OSA patients, who will be divided into two four groups: Control, OPR, CPAP alone and CPAP+OPR. The OPR training in OPR and CPAP+OPR groups will consist of home-based exercises performed for 30-45 minutes per session, once 1-2 session a day, five 3-5 days a week, over a period of three months. The training will be monitored using a strength sensor, and the intensity of the exercises will be adjusted every two weeks month during hospital visits. Both CPAP and CPAP+OPR groups will continue to wear CPAP every night, while the control group will receive monthly sleep hygiene education. The severity of OSA, upper airway space, tongue muscle length/thickness, tongue muscle strength/endurance, sleep quality, and CPAP usage report will be assessed using polysomnography, computed tomography scans, sonography, tongue muscle function tests, sleep quality questionnaires, and CPAP mask pressure at baseline and after three months of treatment.

Expected outcomes：

1. Compared to the group using only CPAP, the CPAP + OPR group will have an increased upper airway space volume after a 3-month follow-up. The upper airway space volume is negatively correlated with CPAP pressure and positively correlated with tongue muscle strength.
2. After 3 months of OPR treatment, the CPAP + OPR group will show an increase in tongue muscle strength, which is negatively correlated with CPAP pressure.
3. After 3 months of OPR treatment, both the OPR group and the CPAP+OPR group showed greater improvements in upper airway muscle function and greater reductions in obstructive sleep apnea severity and clinical symptoms compared to the control group and the CPAP group respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 68 years
* Newly diagnosed with mild to severe pure obstructive sleep apnea based on polysomnography

Exclusion Criteria:

* Severe allergic rhinitis
* Sinusitis with nasal polyps
* Adenoid hypertrophy
* Bilateral tonsillar hypertrophy (Friedman grade ≥ III)
* Lingual tonsil hypertrophy (Friedman grade ≥ III)
* Body Mass Index (BMI) > 40
* Alcohol or drug abuse within the past year
* Pregnancy
* Severe obstructive or restrictive pulmonary diseases
* High-risk cardiovascular diseases during exercise (e.g., angina, myocardial infarction, heart failure, valvular heart disease)
* History of central or peripheral neurological disorders that interfere with exercise prescription
* Musculoskeletal or psychological disorders that interfere with exercise prescription
* Other non-respiratory sleep disorders
* Sleep disorders with concomitant central sleep apnea

Ages: 20 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index | Baseline and 12 weeks post intervention
  The apnea-hypopnea index will be obtained from the overnight Polysomnography (PSG) study. PSG will be performed in the sleep center of National Cheng Kung University Hospital. Less than 5 events/hour indicates normal; AHI between 5-14 events/hour indicates mild Obstructive Sleep Apnea(OSA); AHI between 15-30 events/hour indicates moderate OSA; and AHI more than 30 events/hour indicates severe OSA.

SECONDARY OUTCOMES:
Tongue Muscle Strength | Baseline and 12 weeks post intervention
  The maximal muscle strength of genioglossus muscles using The Iowa Oral Performance Instrument (IOPI) system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA) (kPa)
Tongue Muscle Endurance | Baseline and 12 weeks post intervention
  The endurance of the genioglossus muscles using The Iowa Oral Performance Instrument (IOPI) system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA) (in seconds).
Pharyngeal Airway Volume | Baseline and 12 weeks post intervention
  Computer Tomography (CT) will be performed. The pharyngeal airway volume will be calculated from the hard palate to the epiglottis and the data will be presented in cm^3. The minimum score is 0 and a higher score indicates greater in pharyngeal airway volume.
Cross Section Area on the Tip of Epiglottis | Baseline and 12 weeks post intervention
  Computer Tomography (CT) will be performed. Cross section area on the tip of the epiglottis was measured and the data will be presented in cm^2. The minimum score is 0 and a higher score indicates greater in the cross-sectional area of the region.
Anterior to Posterior Distance on the Tip of the Epiglottis | Baseline and 12 weeks post intervention
  The distance between the anterior and posterior pharyngeal wall on the tip of the epiglottis will be measured and presented in cm. The minimal value will be 0 and the greater value indicates a greater distance between the anterior to posterior in this area.
Lateral Distance on the Tip of Epiglottis | Baseline and 12 weeks post intervention
  The distance between the lateral distance on the tip of the epiglottis will be measured and presented in cm. The minimal value will be 0 and the greater value indicates a greater distance between the lateral wall.
Sleep Quality | Baseline and 12 weeks post intervention
  Sleep quality will be measured using Pittsburgh Sleep Quality Index (PSQI).The total score ranges from 0 to 21 with a higher total score equal to or more than 5 indicating worse sleep quality.
Daytime Sleepiness Level | Baseline and 12 weeks post intervention
  Epworth Sleepiness Score(ESS) will be used to measure the daytime sleepiness of OSA patients. The total score of ESS range from 0-24. A score greater than 10 indicates greater daytime sleepiness.
Tongue Muscle Thickness | Baseline and 12 weeks post intervention
  Sonography will be performed over the participant's neck region to assess the changes in tongue muscle thickness during normal breathing and Müller's maneuver. The data on tongue thickness will be presented in millimeters. A greater value indicates a thicker in tongue.
Median Pressure in Continuous Positive Airway Pressure | 1-week average pre intervention, 1-week average post intervention and 1-month average during intervention for 3 months
  The change in therapeutic CPAP pressure required to maintain airway patency will be assessed using CPAP usage reports. A reduction in required pressure is expected to indicate improved upper airway muscle tone and stability.
Median Usage Hours of Continuous Positive Airway Pressure | 1-week average pre intervention, 1-week average post intervention and 1-month average during intervention for 3 months
  The average number of hours per night that participants use CPAP will be recorded from CPAP usage reports. Greater nightly usage is considered indicative of better compliance and treatment effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hsia Hung, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No